CLINICAL TRIAL: NCT07070583
Title: Impact of Endovascular Treatment of Aorto-iliac Disease on Systemic Hypertension A Pilot Study Impact of Aorto-Iliac Occlusive Disease Treatment on Blood Pressure
Brief Title: Impact of Aorto-Iliac Occlusive Disease Treatment on Blood Pressure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Blood pressure in AIOD
Record Dates: First submitted 2025-06-30; First posted 2025-07-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Aorto Iliac Occlusive Disease; Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stent placement (Other): Patients with an aorto-iliac occlusion will receive a stent, according to standard care
  Interventions: Procedure: Stent placement

INTERVENTIONS:
Procedure: Stent placement — Patients with an aorto-iliac occlusion will receive a stent, according to standard care

SUMMARY:
Hypertension is a major risk factor for a variety of cardiovascular diseases. When hypertension results from increased vascular resistance due to a narrowing of the descending aorta, it can be effectively treated with stenting. More recently, evidence suggest that stenting in more distal parts of the arterial vascular bed is also associated with a reduction in blood pressure. The investigators hypothesize that stenting of occlusions more distal of the descending aorta decreases the central blood pressure and afterload as reflected by NT-proBNP (N-terminal pro-Brain Natriuretic Peptide), a biomarker of intracardiac pressures and predictor of heart failure events. The goal of this pilot study is to prospectively investigate changes in blood pressure after stent placement in the aorto-iliac region.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Singed informed consent
* Chronic occlusion in the infrarenal aorta and/or one or both common iliac arteries
* Total lesion length of ≥30mm
* Clinical indication for treatment of the pathology (Chronic limb threatening ischemia or disabling intermittent claudication not responding to supervised exercise training)

Exclusion Criteria:

* Patient is unable to understand the study requirements and/ or is unwilling to adhere to the follow-up
* Juxtarenal pathology (<2cm below the lowest renal artery)
* Acute occlusion of the target area (Acute Leriche Syndrome)
* Embolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to describe the changes in arterial blood pressures between baseline and 12 months follow-up after endovascular treatment of an occlusion of the infrarenal aorta and/or common iliac arteries. | 12 months

SECONDARY OUTCOMES:
To gather information about the association between cardiac biomarkers (hemoglobin, creatinin, NT-pro-BNP) on blood pressure at 12 months in patients with treatment for an occlusion of the infrarenal aorta and/or common iliac arteries. | 12 months
To determine if treatment of an occlusion of the infrarenal aorta and/or common iliac arteries will change the Pulse Wave Analysis (PWA) Pulse Wave Velocity (PWV) measurements at 12 months, compared to baseline. | 12 months
To investigate if treatment of an occlusion of the infrarenal aorta and/or common iliac arteries will decrease or increase the number of anti-hypertensive medication use at 12 months, compared to baseline. | 12 months

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet